CLINICAL TRIAL: NCT05177965
Title: The Metabolic and Circadian Effects of Shift Work - An Observational Study
Brief Title: The Metabolic and Circadian Effects of Shift Work
Acronym: OPTI-SHIFT
Status: Completed | Type: Observational
Sponsor: Tinh-Hai Collet, MD (Other)
Responsible Party: Sponsor-Investigator, Tinh-Hai Collet, MD, Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: 2021-01088
Record Dates: First submitted 2021-11-18; First posted 2022-01-05 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Shift Work Schedule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Shift workers: Measurements repeated during a series of day shifts and during a series of night shifts
  Interventions: Other: Exposure to shift work

INTERVENTIONS:
Other: Exposure to shift work — Detailed questionnaire adapted from the Standard Shiftwork Index, measured at inclusion

SUMMARY:
In an exploratory observational pilot study, the investigators will focus on the effects of short-term circadian misalignment induced by shift work on multidimensional measurements including glucose excursion, metabolic health, circadian rhythms (measured in vitro and in vivo), sleep/wake cycles and ambient light, eating and activity patterns, well-being and attention.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age 20-50 years
* Working ≥ 80% full-time equivalent over the previous month and during the study
* Working night shifts (i.e. shifts that comprise working hours between 23h and 06h) in rotation with day shifts (i.e. shifts that comprise working hours between 06h and 20h)
* Planned to work at least 3 consecutive night shifts during the study preceded by at least a day off or day shift
* Planned to work at least 3 consecutive day shifts during the study
* Confident use of a smartphone compatible with the study application (iOS, Android) and able to regularly take pictures of consumed food/drinks
* Able to give a fully informed consent and follow the study procedures

Exclusion Criteria:

* Planned or current pregnancy during the study
* Menopausal women
* Major illness or hospitalization over the previous month
* Carries a pacemaker, pump or other medical device that can be disabled by a magnet
* Major mental illness
* Trip to a different time zone (≥ 2-hour time difference) over the previous month or planned during the study
* Enrolled in an interventional clinical trial (potentially interfering with the main outcomes) over the previous month or planned during the study

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Shift workers
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Difference in glucose excursion | Between a series of day shifts and a series night shifts, separated by an interval from 10 days to 3 months
  As measured by Continuous Glucose Monitoring

SECONDARY OUTCOMES:
Difference in fasting glucose | Between a series of day shifts and a series night shifts, separated by an interval from 10 days to 3 months
  As measured by clinical chemistry (mmol/L)
Difference in weight | Between a series of day shifts and a series night shifts, separated by an interval from 10 days to 3 months
  Body weight (Kg)
Difference in waist circumference | Between a series of day shifts and a series night shifts, separated by an interval from 10 days to 3 months
  Waist circumference (cm) assessed with a measuring tape
Difference in lipid profile | Between a series of day shifts and a series night shifts, separated by an interval from 10 days to 3 months
  Total cholesterol, triglycerides, HDL cholesterol, LDL cholesterol measured by clinical chemistry (mmol/L)
Difference in blood hormonal profile | Between a series of day shifts and a series night shifts, separated by an interval from 10 days to 3 months
  Insulin (mIU/L), thyroid-stimulating hormone (mIU/L), cortisol (nmol/L) measured by clinical chemistry
Difference in eating duration | Between a series of day shifts and a series night shifts, separated by an interval from 10 days to 3 months
  Time from the first to last caloric intake over a 24-hour period
Difference in nutrient intake | Between a series of day shifts and a series night shifts, separated by an interval from 10 days to 3 months
  Total calorie and macronutrient intake over a 24-hour period
Difference in systolic and diastolic blood pressure | Between a series of day shifts and a series night shifts, separated by an interval from 10 days to 3 months
  As measured by blood pressure arm cuff
Difference in heart rate variability | Between a series of day shifts and a series night shifts, separated by an interval from 10 days to 3 months
  As measured by wearable sensor
Difference in physical activity | Between a series of day shifts and a series night shifts, separated by an interval from 10 days to 3 months
  As measured by actigraphy and the International Physical Activity Questionnaire
Difference in sleep/wake cycles | Between a series of day shifts and a series night shifts, separated by an interval from 10 days to 3 months
  As measured by actigraphy
Difference in sleep quality | Between a series of day shifts and a series night shifts, separated by an interval from 10 days to 3 months
  As measured by the Pittsburgh Sleep Quality Index (PSQI), score ranges from 0 to 21 points, 0 indicating no difficulty and 21 severe difficulties
Difference in attention and sleepiness | Between a series of day shifts and a series night shifts, separated by an interval from 10 days to 3 months
  As measured by the Sustained Attention to Response Test
Difference in well-being | Between a series of day shifts and a series night shifts, separated by an interval from 10 days to 3 months
  As measured by the World Health Organization-5 questionnaire (WHO-5), score ranges from 0 to 25, 0 indicating worst possible and 25 best possible
Difference in mental health outcomes | Between a series of day shifts and a series night shifts, separated by an interval from 10 days to 3 months
  As measured by the Patient Health Questionnaire-9 (PHQ-9), score ranges from 0 to 27, 0 indicating no depression and 27 severe depression

OTHER OUTCOMES:
Difference in blood metabolomic parameters | Between a series of day shifts and a series night shifts, separated by an interval from 10 days to 3 months
  As measured by high-throughput mass spectrometry metabolomics, semi-quantitative identification of small metabolites involved in carbohydrate, fat, protein, and steroid metabolism
Difference in lipid metabolism | Between a series of day shifts and a series night shifts, separated by an interval from 10 days to 3 months
  As measured by high-throughput mass spectrometry lipidomics
Difference in the exposure to ambient light | Between a series of day shifts and a series night shifts, separated by an interval from 10 days to 3 months
  As measured by wearable spectrometer and the light exposure behaviour assessment (LEBA) questionnaire
Difference in the core body temperature | Between a series of day shifts and a series night shifts, separated by an interval from 10 days to 3 months
  As measured by a wearable skin temperature and heat transfer sensor

CONTACTS AND LOCATIONS:
Overall Officials: Tinh-Hai Collet, MD, Principal Investigator — Geneva University Hospitals, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

REFERENCES:
- [Result] Hartmeyer SL, Phillips NE, Jassil FC, Joris C, Dibner C, Collet TH, Andersen M. Multi-Wearable Approach for Monitoring Diurnal Light Exposure and Body Rhythms in Nightshift Workers. Acta Physiol (Oxf). 2025 Jul;241(7):e70069. doi: 10.1111/apha.70069. PMID 40485643